CLINICAL TRIAL: NCT00844012
Title: Continuous Versus Cyclic Postoperative Use of Low-Dose Combined Oral Contraceptive Belara® for the Treatment of Endometriosis-Related Chronic Pelvic Pain: a Randomized Controlled Trial.
Brief Title: Continuous Postoperative Use of Low-Dose Combined Oral Contraceptivesfor for Endometriosis-Related Chronic Pelvic Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Fulvio Zullo, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01/2009
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-02

CONDITIONS: Endometriosis; Chronic Pelvic Pain
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: Continuous OC (clormadinone acetate plus ethinil-estradiol - Belara®, Grunenthal, Milan, Italy)
- Control (Active Comparator)
  Interventions: Drug: Cyclic OC (clormadinone acetate plus ethinil-estradiol)

INTERVENTIONS:
Drug: Continuous OC (clormadinone acetate plus ethinil-estradiol - Belara®, Grunenthal, Milan, Italy) — Low-dose monophasic OC containing 2.0 mg clormadinone acetate plus 0.03 mg ethinil-estradiol (Belara®, Grunenthal, Milan, Italy) will be administered with a continuous regimen.
  Arms: Experimental group
Drug: Cyclic OC (clormadinone acetate plus ethinil-estradiol) — Low-dose monophasic OC containing 2.0 mg clormadinone acetate plus 0.03 mg ethinil-estradiol (Belara®, Grunenthal, Milan, Italy) will be administered with a cyclic regimen.
  Arms: Control

SUMMARY:
Because ovarian sex steroids fluctuations during the menstrual cycle are implicated in the pathogenesis of the endometriosis-related chronic pelvic pain (CPP), the oral contraceptives (OCs) are used with non-contraceptive indication for this disorder.

To date, OCs are widely used as medical treatment in patients with endometriosis, in addition, they are recently experimented as post-surgical therapy. Traditional cyclic regimen, with 21 days of active pills with 7 days of placebo or suspension, is usually adopted. Furthermore, recent studies suggested that long-term continuous OCs use can be effective in the postoperative period both as second- and third- line treatments after cyclic regimen failure. In these studies a combined treatment with ethinilestradiol (0.02 mg) plus desogestrel (0.15 mg) were used and compared with baseline or ciproterone acetate.

A recent study showed a deeper ovarian and endometrial suppression with continuous OCs in comparison with cyclic OCs, providing a physiological rationale for continuous OCs use for noncontraceptive indications. Furthermore, to date, no study compared post-operative continuous versus cyclic OCs in patients with endometriosis-related CPP.

DETAILED DESCRIPTION:
Premenopausal women with endometriosis-related CPP scheduled for laparoscopic surgery to our Academic Department of Gynecology will be consecutively enrolled. Subjects with hystologically confirmed endometriosis at laparoscopy (stage I-IV of the American Society Reproductive Medicine), a subjective severity of pelvic pain by using a visual analogue scale (VAS 1-100) of at least 70, and without immediate desire of pregnancy will be enrolled.

Briefly, all patients will undergo conservative laparoscopic surgery for endometriosis. Thereafter, a low-dose monophasic OC containing 2.0 mg clormadinone acetate plus 0.03 mg ethinil-estradiol (Belara®, Grunenthal, Milan, Italy) will be administered. Patients from the experimental group will be treated with a continuous regimen, while patients from the control group will receive the OC with a cyclic regimen consisting of 21 days of active pills with 7 days of placebo. The drug and the placebo will be similar and will be labelled according to the subject number. For the overall study-period, operators and patients will be blind to the treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal state
* Endometriosis-related chronic pelvic pain
* Hystologically confirmed endometriosis at laparoscopy
* Subjective severity of pelvic pain by using a visual analogue scale of at least 70
* No immediate desire of pregnancy

Exclusion Criteria:

* Age ≤18 or ≥ 40
* Previous use of drugs for treating CPP (wash-out period of 3 months), with exclusion of non-steroidal anti-inflammatory drugs
* Contraindication to estro-progestin compounds
* Major medical diseases
* Psychiatric disorders
* Pelvic inflammatory disease
* Adnexal patologies
* Unability to complete the daily diary
* History of alcohol or other drugs abuse

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Recurrence of pelvic pain | 12 months

SECONDARY OUTCOMES:
Metabolic effects | 12 months
Ovarian effects | 12 months
Endometrial effects | 12 months
Bleedings characteristics | 12 months
Protocol adherence | 12 months
Satisfaction rate | 12 months
Adverse events | 12 months
Effects on cognitive function and mood | 12 months
Quality of life | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Catanzaro, Italy, Catanzaro, Italy